CLINICAL TRIAL: NCT03787134
Title: Oscillatory Contributions to Working Memory and Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-0500; A538900 (Other: UW Madison); SMPH\PSYCHIATRY\PSYCHIATRY (Other: UW Madison); 2R01MH095984-06 (NIH); Protocol Version 8/11/2022 (Other: UW Madison)
Record Dates: First submitted 2018-12-14; First posted 2018-12-26 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Young Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2016-0500-Healthy YoungAdults (Experimental): working memory and attention
  Interventions: Behavioral: working memory and attention

INTERVENTIONS:
Behavioral: working memory and attention — Behavioral tests of working memory and attention

SUMMARY:
The objectives are articulated in the proposal's specific aims:

Aim 1: To test the hypothesis that the cognitive control of unattended memory items (UMI) is implemented by the same frontoparietal mechanisms that control spatial and nonspatial attention.

Aim 2: To test the hypothesis that the selection of visual stimuli, whether from the environment or from WM, is accomplished, in part, by the hijacking of low-frequency oscillatory dynamics that are fundamental to the waking-state physiology of the corticothalamic circuitry of the visual system.

Aim 3: To test the hypothesis that the function of context binding contributes to delay-period activity of the posterior parietal cortex (PPC).

DETAILED DESCRIPTION:
4.2.a Narrative Study Description There are 11 distinct experiments proposed, and each is described in turn. Experiment 1.a.: Unconfounding cognitive state from the passage of time for UMI reactivation This experiment entails recording the EEG, and delivering spTMS, while healthy young adult subjects perform two types of WM trials: dual serial retrocuing (DSR) trials and single-retrocue trials. DSR trials begin with the presentation of two items (drawn from categories face, motion, word), followed by an initial Delay 1.1, then Cue 1 indicating which of the two will be probed by the first memory probe. After Probe 1, Cue 2 indicates which item will be tested by Probe 2. Both trial types will feature 3 types of probe: match (50% of trials); nonmatch/same-category (drawn from same category as retrocued sample, 30% of trials); and nonmatch/lure (probe is the uncued item, 20% of trials. spTMS will also be delivered, unpredictably on half of the delay periods, to IPS2. Prospective power analysis, using the results from PMC 5221753 (and taking into account that Exp. 1.a., unlike PMC 5221753, will use a repeated measures design), indicates that 360 trials per subject, and 12 subjects, are required to achieve 80% power for the critical behavioral comparison, which is the comparative influence of spTMS on the FAR to nonmatch/lure probes for dual serial- vs. single-retrocue trials, assessed with the contrast [(FAR nonmatch/lure, dual - FARnonmatch/same-category, dual) - (FAR nonmatch/lure, single - FARnonmatch/same-category, single)]. (To balance the number of match and nonmatch probes, there will be a total of 720 trials per subject.) Each subject will participate in two 2.5-hr experimental sessions. (Allowing for 15% attrition inflates the target n from 12 to 14.)

Exp. 2.a. spTMS/EEG of the frontoparietal salience map. Study PMC 4893488 used n of 17 to achieve reliable single-trial regression results, which are least-powered analyses planned with this dataset; 18 subjects will allow for same number of subjects per targeted hemisphere. From the perspective of counterbalancing order of region targeted with spTMS, 12 subjects would be needed (2 hemispheres * 6 possible orders); once the 12 counterbalancing cells have been filled, the remaining 6 subjects will be selected two-at-a-time, and assigned the same randomly selected order-of-region, one to each hemisphere). (Allowing for 15% attrition inflates the target n from 18 to 21.)

Exp. 2.b. 1 Hz rTMS of the frontoparietal salience map. Study PMC 5725229 recruited 27 subjects, based on its own power analysis based on the literature, to use a rTMS procedure comparable to what Exp. 2.b. will use to disrupt the function of PFC, one of the regions that will be targeted in this study. Because several previous studies using TMS to study attentional selection have found evidence of hemispheric asymmetries in the control of spatial attention, 27 subjects per hemisphere to be targeted will be recruited, yielding a total of 54. (Allowing for 15% attrition inflates the target n from 54 to 62.)

Exp. 2.c.1 Hz rTMS of FEF and IFJ. Considerations are identical to those for Exp. 2.b.

Experiment 3.a. Studying alpha-band dynamics of spatial and temporal attention with EEG.

Study PMC 4500270 found reliable effects of temporal prediction-related frequency-shifting in the alpha band with 15 subjects. Sixteen (16) subjects will be recruited in order to achieve equal counterbalancing. (Allowing for 15% attrition inflates the target n from 16 to 18.)

Exp. 4.a. Strategic control of alpha-band dynamics for perceptually unchallenging visual selection.

Considerations are identical to those for Exp. 3.a.

Exp. 4.b. Strategic control of alpha-band dynamics for selection in visual WM. Considerations are identical to those for Exp. 3.a.

Experiment 5 (addressing Aim 3). Testing WM storage vs. context binding accounts of the CDA Power analyses, carried out with resampling of simulated data derived from the preliminary results of this study, indicate that 36 subjects are needed for 90% power to detect a load effect (i.e., CDA for 3C trials > CDA for 1C trials). (Allowing for 15% attrition inflates the target n from 36 to 41.)

Experiment 6 (addressing Aim 3). Varying the domain of context. Considerations are identical to those for Exp. 5.

ELIGIBILITY:
Inclusion Criteria:

* Age of # 18 <36. - Right-handed.
* Be in good health determined by the investigator on basis of medical history, physical and neurological exam; for "EEG-only" sessions no physical or neurological exams will be performed;
* Female subjects must be two years past menopause, surgically sterile or practicing a medically acceptable method of birth control (does not apply to "EEG-only" sessions);
* Female subjects must not be pregnant.
* Able to understand and speak English.
* Able to provide written consent prior to admission

Exclusion Criteria:

* History of epilepsy, stroke, brain surgery, cranial metal implants, structural brain lesion, devices that may be affected by TMS or tCS(pacemaker, medication pump, cochlear implant, implanted brain stimulator); - Women who are breast-feeding (self report)*;
* History of head trauma with loss of consciousness for greater than 5 minutes;
* Any history of seizures;
* Any family history of seizures*;
* Diabetes requiring insulin treatment*;
* A serious heart disorder or subjects who have had a heart attack within the last 3 months;
* Subjects who meet DSM-IV criteria for alcohol /drug abuse problems within the last six months;
* Any current Axis I or II diagnoses or past Axis I diagnoses;
* Required use of medication that affects CNS function;
* A subject with metallic implants, such as prostheses, shrapnel or aneurysm clip-S, or persons with electronic implants, such as cardiac pacemakers. The magnetic field generated by the MR machine can cause a displacement or malfunctioning of these devices*;
* The female subject who is pregnant or planning to become pregnant; or a female subject of child-bearing potential who is not practicing a medically acceptable form of birth control*;
* The subject has had a diagnosis of cancer in the past 3 years and/or has active neoplastic disease;
* The investigator anticipates that the subject will be unable to comply with the protocol.
* Prohibited Concomitant Treatment: Any investigational medication; antipsychotic, antidepressant; or ECT; Other psychotropic medications including sedative hypnotics (excluding chloral hydrate zaleplon); sumatriptan (and similar agents); anxiolytics and herbals (e.g., St. John's Wort, Kava Kava); an introduction or change in intensity of psychotherapy; any nonpsychopharmacologic drug with psychotropic effects (e.g., antihistamines, beta blockers).
* Colorblindness
* Poor or Uncorrected Vision
* History of fainting/syncope

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fulvio JM, Postle BR. Cognitive Control, Not Time, Determines the Status of Items in Working Memory. J Cogn. 2020 Apr 9;3(1):8. doi: 10.5334/joc.98. PMID 32292872
- [Result] Pietrelli M, Samaha J, Postle BR. Spectral Distribution Dynamics across Different Attentional Priority States. J Neurosci. 2022 May 11;42(19):4026-4041. doi: 10.1523/JNEUROSCI.2318-21.2022. Epub 2022 Apr 6. PMID 35387871
- [Result] Wan Q, Cai Y, Samaha J, Postle BR. Tracking stimulus representation across a 2-back visual working memory task. R Soc Open Sci. 2020 Aug 5;7(8):190228. doi: 10.1098/rsos.190228. eCollection 2020 Aug. PMID 32968489
- [Result] Cai Y, Fulvio JM, Samaha J, Postle BR. Context Binding in Visual Working Memory Is Reflected in Bilateral Event-Related Potentials, But Not in Contralateral Delay Activity. eNeuro. 2022 Nov 9;9(6):ENEURO.0207-22.2022. doi: 10.1523/ENEURO.0207-22.2022. Print 2022 Nov-Dec. PMID 36265905

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-study 1: Working memory task with categorical stimuli of faces, words, and dot motion, involving delayed recognition responses; EEG recorded and single-pulse TMS applied intermittently during delay periods. n = 12
- Sub-study 2: 2-back working memory task with EEG recorded involving 'match'/'non-match' responses; n = 30
- Sub-study 3: Posner-style visual cueing task involving orientation judgments; n = 19
- Sub-study 4: Visual working memory task with three categories of stimuli: orientations, luminances, colors, and involving 'match'/'non-match' responses with EEG recorded; n = 28
- Sub-study 5: Dual task with delayed recall of orientation (working memory) and visual discrimination of orientation during the delay period (perception) with EEG recorded; n = 25
- Sub-study 6: Visual working memory task with delayed recognition responses ('match'/'non-match') of object color or orientation with EEG recorded; n = 56
- Sub-study 7: Delayed-recall of orientation working memory task with EEG recorded; n = 14
Period: Overall Study
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Started | 12 | 30 | 19 | 28 | 25 | 56 | 14
Outcome 1 - Behavioral Accuracy (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 12 | 30 | 19 | 0 | 25 | 0 | 0
Outcome 2 - Reaction Time (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 12 | 30 | 19 | 0 | 25 | 56 | 0
Outcome 3 - Multivariate Pattern Classification of EEG (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 12 | 0 | 0 | 0 | 0 | 0 | 0
Outcome 4 - Component Loadings (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 12 | 0 | 0 | 0 | 0 | 0 | 0
Outcome 9 - Alpha Band Power (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 0 | 0 | 19 | 0 | 0 | 0 | 0
Outcome 12 - Behavioral Accuracy (Mean Recall Error) (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 0 | 0 | 0 | 0 | 0 | 0 | 14
Outcome 17 - Amplitude of CDA (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 0 | 0 | 0 | 28 | 0 | 56 | 0
Outcome 18 - IEM (Number of Participants who contributed data for outcome by experimental design, not all sub-studies were designed to collect data for all outcomes.) | 0 | 30 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 30 | 19 | 28 | 25 | 56 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7 | Total
Number analyzed (Participants) | 12 | 30 | 19 | 28 | 25 | 56 | 14 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 30 | 19 | 28 | 25 | 56 | 14 | 184
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristic of 'female' and 'male' is based on voluntary participant reports. In some instances, participants have opted not to disclose this information and as a result, the number analyzed in a particular sub-study will be different from the overall total enrolled.
  Participants
    number analyzed (Participants) | 12 | 30 | 19 | 27 | 25 | 43 | 14 | 170
    Female | 5 | 19 | 11 | 19 | 12 | 32 | 11 | 109
    Male | 7 | 11 | 8 | 8 | 13 | 11 | 3 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 12 | 28 | 19 | 25 | 20 | 54 | 14 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 12 | 7 | 22 | 5 | 53 | 14 | 115
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
  White | 10 | 12 | 12 | 4 | 16 | 0 | 0 | 54
  More than one race | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 4 | 3 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 12 | 30 | 19 | 28 | 25 | 56 | 14 | 184

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Accuracy: Sub-study 1
Description: Mean percentage of correct recognition responses - indicates the percentage of trials, on average, participants correctly identified a test stimulus as a match or non-match to an item in working memory. The primary task completed by this group was a dual-serial recognition (DSR) task which involved two responses on each trial. The secondary (control) task was a single recognition (SR) task which involved one response on each trial. The two tasks were interleaved, so all participants completed them in succession throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded and single-pulse TMS applied intermittently during delay periods. Sub-study 1 participants only.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Sub-study 1: Working memory task with categorical stimuli of faces, words, and dot motion, involving delayed recognition responses
Arm/Group | Sub-study 1
Number analyzed (Participants) | 12
percentage of correct responses
  DSR task | 86.3 (9.2)
  SR task | 87.1 (10.3)

2. Primary Outcome: Behavioral Accuracy: Sub-study 2
Description: Mean percentage of correct recognition responses - indicates the percentage of trials, on average, participants correctly identified a test stimulus as a match or non-match to an item in working memory. The primary task completed by this group of participants was a two-back recognition task, in which participants indicated whether the current stimulus was a match or non-match to the stimulus shown two items ago (completed during the first half of the measured time frame); the second task was a delayed recognition task in which participants indicated whether the current stimulus was a match or non-match to a stimulus shown 1750 ms prior (completed during the second half of the measured time frame).
Time Frame: 3 hours
Population: EEG recorded; sub-study 2 participants only
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Sub-study 2: 2-back working memory task with secondary delayed recognition task involving 'match'/'non-match' responses
Arm/Group | Sub-study 2
Number analyzed (Participants) | 30
percentage of correct responses
  2-back task | 85.7 (6.0)
  delayed recognition task | 78.5 (7.0)

3. Primary Outcome: Behavioral Accuracy: Sub-study 3
Description: Mean percentage of correct recognition responses - indicates the percentage of trials, on average, participants correctly identified a test stimulus as a match or non-match to an item in working memory. The primary task results were based on validly cued trials in which the cue indicated the to-be-tested location, whereas the second task results were based on the invalidly cued trials in which the cue indicated a location that was not the to-be-tested location. These task conditions were intermixed throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded; sub-study 3 participants only
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Sub-study 3: Posner-style visual cueing task involving orientation judgments
Arm/Group | Sub-study 3
Number analyzed (Participants) | 19
percentage of correct responses
  Valid cueing | 72 (10)
  Invalid cueing | 67 (9)

4. Primary Outcome: Behavioral Accuracy: Sub-study 5
Description: Mean percentage of correct recognition responses - indicates the percentage of trials, on average, participants correctly identified a test stimulus as a match or non-match to an item in working memory. The primary task results were based on the accuracy of discrimination on 'congruent' trials in which the working memory item and the perceptual discrimination stimulus were identical in orientation; the secondary task results were based on the accuracy of discrimination on 'incongruent' trials. The two task types were intermixed throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded; sub-study 5 participants only
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Sub-study 5: Dual task with delayed recall of orientation (working memory) and visual discrimination of orientation during the delay period (perception).
Arm/Group | Sub-study 5
Number analyzed (Participants) | 25
percentage of correct responses
  Congruent trials | 86.5 (2.1)
  Incongruent trials | 86 (2)

5. Primary Outcome: Behavioral Accuracy: Sub-study 7
Description: Mean error (in degrees). On each trial, participants must memorize three object orientations (e.g. 10, 40, and 75 degrees) that are shown at different locations in succession on a computer screen. Several seconds later, the participant is given a cue/indicator about which of the orientations they will need to recall (i.e., reproduce) during the trial's test phase. After another brief delay, a line is shown on the screen and the participant must rotate it with the mouse to match the orientation in memory. This occurred in two task conditions: the 'overlap' condition in which two memory items were shown at the same location on the screen; and the 'non-overlap' condition, in which all items were presented at different locations on the screen. The 'overlap' task was carried out in the first half of the measured time frame; the 'non-overlap' task was carried out in the second half. Large errors (big differences between the reported and displayed orientation) indicate worse memory accuracy.
Time Frame: 4 hours
Population: EEG recorded; sub-study 7 participants only
Measure: Mean (Standard Deviation); unit: degrees (of orientation)
Groups:
- Sub-study 7: Delayed-recall of orientation working memory task.
Arm/Group | Sub-study 7
Number analyzed (Participants) | 14
degrees (of orientation)
  Overlap task | 11.96 (3.12)
  Non-overlap task | 13.12 (3.2)

6. Primary Outcome: Reaction Time: Sub-study 1
Description: The time, measured in milliseconds, that it took a subject to lock in their response via keyboard button press on each trial. The primary task completed by this group was a dual-serial recognition (DSR) task which involved two responses on each trial. The secondary (control) task was a single recognition (SR) task which involved one response on each trial. The two tasks were interleaved, so all participants completed them in succession throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded and single-pulse TMS applied intermittently during delay periods. Sub-study 1 participants only
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sub-study 1
Number analyzed (Participants) | 12
milliseconds
  DSR task | 811 (130)
  SR task | 823 (123)

7. Primary Outcome: Reaction Time: Sub-study 2
Description: The average time, measured in milliseconds, that it took a subject to lock in their response via mouse button click on each trial. The primary task completed by this group of participants was a two-back recognition task, in which participants indicated whether the current stimulus was a match or non-match to the stimulus shown two items ago (completed during the first half of the measured time frame); the second task was a delayed recognition task in which participants indicated whether the current stimulus was a match or non-match to a stimulus shown 1750 ms prior (completed during the second half of the measured time frame).
Time Frame: 3 hours
Population: EEG recorded; sub-study 2 participants only
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Sub-study 2: 2-back working memory task with EEG recorded involving 'match'/'non-match' responses.
Arm/Group | Sub-study 2
Number analyzed (Participants) | 30
milliseconds
  2-back task | 850 (210)
  delayed recognition task | 660 (120)

8. Primary Outcome: Reaction Time: Sub-study 3
Description: The average time, measured in milliseconds, that it took a subject to lock in their response via keyboard button press on each trial. The primary task results were based on validly cued trials in which the cue indicated the to-be-tested location, whereas the second task results were based on the invalidly cued trials in which the cue indicated a location that was not the to-be-tested location. These task conditions were intermixed throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded; sub-study 3 participants only
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sub-study 3
Number analyzed (Participants) | 19
milliseconds
  Valid cueing | 1004 (309)
  Invalid cueing | 1070 (296)

9. Primary Outcome: Reaction Time: Sub-study 5
Description: The average time, measured in milliseconds, that it took a subject to lock in their response via keyboard button press on each trial. The primary task results were based on the accuracy of discrimination on 'congruent' trials in which the working memory item and the perceptual discrimination stimulus were identical in orientation; the secondary task results were based on the accuracy of discrimination on 'incongruent' trials. The two task types were intermixed throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded; sub-study 5 participants only
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sub-study 5
Number analyzed (Participants) | 25
milliseconds
  Congruent trials | 970 (110)
  Incongruent trials | 990 (140)

10. Primary Outcome: Reaction Time: Sub-study 6
Description: The average time, measured in milliseconds, that it took a subject to lock in their response via keyboard button press on each trial. The primary task was a 'set size 2' task in which participants had to maintain two items in working memory; the secondary task was a 'set size 1' task in which participants maintained one item in working memory. These tasks were intermixed throughout the measured time frame.
Time Frame: 3 hours
Population: EEG recorded; sub-study 6 participants only
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Sub-study 6: Visual working memory task with delayed recognition responses ('match'/'non-match') of object color or orientation.
Arm/Group | Sub-study 6
Number analyzed (Participants) | 56
milliseconds
  Memory set size 2 | 750 (85)
  Memory set size 1 | 675 (80)

11. Primary Outcome: Multivariate Pattern Classification of EEG Data: Sub-study 1
Description: Multivariate pattern classification is a machine learning method that assesses the neural representation of stimulus information in electroencephalographic (EEG) signal (i.e., to "decode" the signal). The outcome measure is decoding performance. When a decoder performs well (here, greater than 0.5), the EEG signal contains information consistent with the representation of the stimulus at that point in the trial; when it performs poorly (here, less than or equal to 0.5), there is no evidence for stimulus representation at that time. Reported here is average classifier accuracy (expressed as area under the curve) in decoding a memory item's representation during the memory period for the different task conditions: when the item was cued or uncued and when transcranial magnetic stimulation (TMS) was delivered or not. The data used come from the full measured time frame.
Time Frame: 3 hours
Population: EEG recorded and single-pulse TMS applied intermittently during delay periods. Sub-study 1 participants only.
Measure: Mean (Standard Error); unit: probability of distinguishing stimuli
Arm/Group | Sub-study 1
Number analyzed (Participants) | 12
probability of distinguishing stimuli
  Item cued + TMS delivered | .55 (.05)
  Item uncued + TMS delivered | .54 (.05)
  Item cued + TMS not delivered | .52 (.1)
  Item uncued + TMS not delivered | .49 (.1)

12. Primary Outcome: Multivariate Inverted Encoding Modeling (IEM) Reconstruction: Sub-study 2
Description: Each EEG electrode's signal was construed as a weighted sum of responses from six channels tuned to specific stimulus orientations in the study. Data from the delayed recognition task were regressed onto this basis set to obtain a weight matrix characterizing the contribution of each channel to each electrode's response. The weight matrix was then inverted to derive the reconstructed representation of stimulus orientation during the delay period of the primary 2-back task data. Reported is the group-level slope (in arbitrary units) of the reconstruction of the cued and uncued memory items during the delay period, serving as a memory strength index/score ranging from -1:+1. Larger slope magnitudes indicate stronger memory representations. Negative values imply that the memory representation was a modified ('flipped') version of the representation held when the stimulus was first presented; positive values indicate direct resemblance to when the stimulus was first presented.
Time Frame: 4 hours
Population: EEG recorded; sub-study 2 participants only
Measure: Number; unit: arbitrary units
Arm/Group | Sub-study 2
Number analyzed (Participants) | 30
arbitrary units
  cued memory item reconstruction | -0.0108
  uncued memory item reconstruction | 0.0033
Statistical Analysis 1: Comparison: Sub-study 2; cued memory item reconstruction - test of reconstruction strength against 0; Test type: Superiority; p = .335, t-test, 2 sided
Statistical Analysis 2: Comparison: Sub-study 2; uncued memory item reconstruction - test of reconstruction strength against 0; Test type: Superiority; p = .016, t-test, 2 sided

13. Primary Outcome: Transcranial Magnetic Stimulation (TMS) Effects on EEG Data Component Strengths: Sub-study 1
Description: The spatially distributed phase coupling extraction (SPACE) decomposition method was used to identify discrete neural rhythms ('components') giving rise to the EEG signal. The strength of identified components at each time point (epoch) in the trial provides a measure of activity, ranging from 0 (absent/inactive) to a positive value (present/active). Strengths were used to address the question of whether single pulse TMS evokes new neural rhythms that weren't active before the pulse or modulates existing rhythms. If new rhythms are evoked, a greater percentage of trials with negligible (~0) strengths prior to TMS that increase after TMS compared to trials without TMS should be observed. Reported are the percentage of trials with this pattern for the posterior beta, posterior alpha, and posterior theta identified components for trials with and without TMS and TMS. Data from the full session were used.
Time Frame: 3 hours
Population: EEG recorded and single-pulse TMS applied intermittently during delay periods; sub-study 1 participants only
Measure: Number; unit: percentage of epochs
Units Other Than Participants: trial epochs
Arm/Group | Sub-study 1
Number analyzed (Participants) | 12
Number analyzed (trial epochs) | 2160
percentage of epochs
  TMS delivered posterior beta: number analyzed (trial epochs) | 360
  TMS delivered posterior beta | 4.57
  TMS not delivered posterior beta: number analyzed (trial epochs) | 360
  TMS not delivered posterior beta | 4.5
  TMS delivered posterior alpha: number analyzed (trial epochs) | 360
  TMS delivered posterior alpha | 40.12
  TMS not delivered posterior alpha: number analyzed (trial epochs) | 360
  TMS not delivered posterior alpha | 40.45
  TMS delivered posterior theta: number analyzed (trial epochs) | 360
  TMS delivered posterior theta | 46.33
  TMS not delivered posterior theta: number analyzed (trial epochs) | 360
  TMS not delivered posterior theta | 45.5

14. Primary Outcome: Alpha Band Power as a Function of Location Relevance in Working Memory: Sub-study 3
Description: Neural activity is comprised of rhythmic activity and aperiodic activity. Alpha rhythmic activity plays important roles in supporting working memory performance and varies according to task demands. EEG data were decomposed into alpha periodic and aperiodic components in order to isolate the alpha frequency band power (8-14 Hz). Participants' task was to make judgments about memorized items shown above, below, left, and right of a central viewing point on the screen. To assess the effects of spatial memory cueing on decomposed alpha, electrodes that showed alpha modulation selective to the four memory locations were first identified. Then, the alpha power in those electrodes was compared as a function of whether the location was attended, unattended, or irrelevant on a particular trial. This was done for two epochs: during the memory delay (350 - 850 ms after sample) and target presentation (850 - 1350 ms after sample). Data from the full session was used for this analysis.
Time Frame: 4 hours
Population: EEG recorded; Sub-study 3 participants only
Measure: Mean (Standard Deviation); unit: microvolts squared / Hz
Arm/Group | Sub-study 3
Number analyzed (Participants) | 19
microvolts squared / Hz
  attended location - memory delay | 6.16 (.24)
  unattended location - memory delay | 6.19 (.24)
  irrelevant location - memory delay | 6.2 (.24)
  attended location - target presentation | 5.83 (.19)
  unattended location - target presentation | 6.05 (.2)
  irrelevant location - target presentation | 6.02 (.2)

15. Primary Outcome: The Amplitude of Contralateral Delay Activity (CDA): Sub-study 4
Description: The CDA is an event-related potential (ERP) derived from posterior electrodes that tracks the amount of information held in working memory, and may also be sensitive to context-binding demands. It becomes more negative with increasing memory load. The CDA was computed from the EEG by averaging the voltage across trials to generate signals that were contralateral or ipsilateral to the memory cue. The "difference wave" was computed by subtracting the ipsilateral signals from contralateral signals. The amplitude of the CDA is reported for two conditions: the large set size tracked participants' CDA when the memory set was homogenous - comprised of multiple items from the same stimulus category thus all were cued; the small set size analyses tracked participants' performance when the memory set was heterogenous - comprised of items from multiple stimulus categories, with only one category being cued for the target response. Data from the full session was used in this analysis.
Time Frame: 4 hours
Population: with EEG recorded; Sub-study 4 participants only
Measure: Mean (Standard Error); unit: microvolts
Groups:
- Sub-study 4: Visual working memory task with three categories of stimuli: orientations, luminances, colors, and involving 'match'/'non-match' responses.
Arm/Group | Sub-study 4
Number analyzed (Participants) | 28
microvolts
  Small set size | .25 (.12)
  Large set size | .2 (.1)

16. Primary Outcome: The Amplitude of the "Contralateral Delay Activity" (CDA): Sub-study 6
Description: The CDA is an event-related potential (ERP) derived from posterior electrodes that tracks the amount of information held in working memory, and may also be sensitive to context-binding demands. It becomes more negative with increasing memory load. The CDA was computed from the EEG by averaging the voltage across trials to generate signals that were contralateral or ipsilateral to the memory cue. The "difference wave" was computed by subtracting the ipsilateral signals from contralateral signals. The amplitude of the CDA is reported for two conditions: The large set size tracked participants' CDA when the memory set was comprised of two target features; the small set size analyses tracked participants' performance when the memory set was comprised of one target feature. Data from the full session was used in this analysis.
Time Frame: 4 hours
Population: EEG recorded; sub-study 6 participants only
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Sub-study 6
Number analyzed (Participants) | 56
microvolts
  Small set size | .6 (.05)
  Large set size | .75 (.1)

17. Primary Outcome: Experiment 2.a. The Amplitude of Multivariate Inverted Encoding Model-reconstructions of Stimulus Location, Derived From the Transcranial Magnetic Stimulation-evoked Response
Description: Multivariate inverted encoding modeling will be used to reconstruct the representation of stimulus locations from the electroencephalography data, and the strength of the representation will be compared across three stimulus conditions. Note that this method entails analysis of the broadband electroencephalographic signal (bandpass filtered from 1-100Hz) in each of two formats: time domain, and spectrally transformed. The spectrally transformed analysis does not entail the separate analysis of discrete functionally defined frequency bands (e.g., alpha, beta, etc.). Rather, spectral power values at every integer frequency from 2 to 20 Hz and at every other integer frequency from 22 to 50 Hz, yielding 34 frequencies per channel, are used as features in the analysis.
Time Frame: 5 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Experiment 2.a. Spatially Distributed Phase Coupling Extraction-identified Components of the Transcranial Magnetic Stimulation-evoked Electroencephalography Signal
Description: Spatially distributed phase coupling extraction-identified components of the transcranial magnetic stimulation-evoked electroencephalography signal will indicate whether the unattended memory item reactivation effect is carried by a de novo component in the electroencephalographic signal, or by a change in the power of one or more components that were present in the signal prior to the delivery of transcranial magnetic stimulation. Note that this method entails analysis of a spectral transformation of the broadband electroencephalographic signal that does not entail the separate analysis of discrete functionally defined frequency bands (e.g., alpha, beta, etc.) Rather, spectral power values at every integer frequency from 2 to 20 Hz and every other integer from frequency from 22 to 30 Hz - yielding 24 frequencies per channel - are entered into the analysis. No a priori assumptions are made about the frequency composition of components that the method will identify.
Time Frame: 5 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Experiment 2.a. Correlation of the Amplitude of Multivariate Inverted Encoding Model-reconstructions of the Location of the Unattended Memory Item With Alpha Band Power.
Description: Correlation of the amplitude of multivariate inverted encoding model-reconstructions of the location of the unattended memory item, derived from the transcranial magnetic stimulation-evoked response, with alpha band power when targeting occipital cortex.
Time Frame: 5 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Experiment 2.a. Correlation of the Amplitude of Multivariate Inverted Encoding Model-reconstructions of the Location of the Unattended Memory Item With Beta-band Power
Description: Correlation of the amplitude of multivariate inverted encoding model-reconstructions of the location of the unattended memory item, derived from the transcranial magnetic stimulation-evoked response, with beta-band power when targeting the intraparietal sulcus.
Time Frame: 5 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Experiment 3.a. Frequency in the Alpha Band of the EEG as a Function of Retinotopic Location
Description: Frequency in the alpha band of the EEG as a function of retinotopic location
Time Frame: 4 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Experiment 3.a. Spatially Distributed Phase Coupling Extraction-identified Components of the Electroencephalography Signal From Signals Corresponding to the Attended Location
Description: Spatially distributed phase coupling extraction-identified components of the electroencephalography signal from signals corresponding to the attended location to assess whether expectation-related shifts in alpha-band frequency are produced by a change in the frequency of one oscillator or by a change in the relative power of multiple oscillators.
Time Frame: 4 hours
Population: No data were collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Experiment 4.a. Reaction Time Assess as Latency to Press Response Button After Onset of Critical Stimulus.
Description: Reaction time assess as latency to press response button after onset of critical stimulus.
Time Frame: 4 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Primary Outcome: Experiment 4.a. Power in the Alpha Band of the EEG as a Function of Retinotopic Location
Description: Power in the alpha band of the EEG as a function of retinotopic location
Time Frame: 4 hours
Population: data were not collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Primary Outcome: Experiment 4.a. Frequency in the Alpha Band of the EEG as a Function of Retinotopic Location
Description: Frequency in the alpha band of the EEG as a function of retinotopic location
Time Frame: 4 hours
Population: data were not collected for this outcome measure.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Experiment 4.a. Spatially Distributed Phase Coupling Extraction-identified Alpha-band Components of the Electroencephalography Signal From Signals Corresponding to the Attended Location
Description: as for outcome 22
Time Frame: 4 hours
Population: data were not collected for this outcome measure
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Experiment 6. Multivariate Inverted Encoding Modeling of the EEG Signal to Determine Whether or Not Contextual Information is Carried in This Signal
Description: Multivariate inverted encoding modeling of the EEG signal to determine whether or not contextual information is carried in this signal. Note that this method entails analysis of the broadband electroencephalographic signal (bandpass filtered from 1-100Hz) in each of two formats: time domain, and spectrally transformed. The spectrally transformed analysis does not entail the separate analysis of discrete functionally defined frequency bands (e.g., alpha, beta, etc.). Rather, spectral power values at every integer frequency from 2 to 20 Hz and at every other integer frequency from 22 to 50 Hz - yielding 34 frequencies per channel -- are used as features in the analysis.
Time Frame: 4 hours
Population: data were not collected for this outcome measure
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: While participant was taking part in the experiment up to 4 hours.
Arm/Group | Sub-study 1 | Sub-study 2 | Sub-study 3 | Sub-study 4 | Sub-study 5 | Sub-study 6 | Sub-study 7
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/30 | 0/19 | 0/28 | 0/25 | 0/56 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/30 | 0/19 | 0/28 | 0/25 | 0/56 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/30 | 0/19 | 0/28 | 0/25 | 0/56 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03787134/Prot_000.pdf